CLINICAL TRIAL: NCT06046755
Title: Evaluation of Changes in the Methylome and Prognosis of Obesity-related Breast Cancer After Nutritional Intervention-induced Weight Loss During the Oncological Treatment
Brief Title: Nutritional Intervention-induced Weight Loss During the Oncological Treatment of Obesity-related Breast Cancer
Acronym: NUTOBREST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Hospital Arquitecto Marcide (Other)
Responsible Party: Principal Investigator, Ana Belén Crujeiras Martínez, Senior Researcher, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/293
Record Dates: First submitted 2023-07-21; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Obesity; Weight Change, Body; Epigenetic Disorder
Keywords: Breast cancer; Obesity; Body composition; Adipose tissue; Weight loss; Ketogenic diet; Group Educational Intervention; DNA methylation; Hormonal adjuvance
MeSH Terms: conditions — Breast Neoplasms; Obesity; Body Weight Changes; Weight Loss

STUDY DESIGN:
Intervention Model Description: Postmenopausal women (n=130) diagnosed with primary, histologically confirmed, incident postmenopausal breast cancer and with 50-70 years at diagnosis will be recruited. A group of 60 breast cancer patients with obesity (BMI≥30) will be invited to follow a weight loss treatment based on a 4 months-energy restriction-ketogenic intervention arm or a behavioural group intervention. Those groups will be compared with a non-intervention control arm of with 30 breast cancer with obesity and 30 normal weight women.
  On the other hand, a group of 90 tumor-free postmenopausal women (50-17 years) will be recruited in the Endocrinology and Nutrition Service of reference hospitals where 30 women will have a normal weight and the other 60 will be women with obesity. These last women will be subjected to a 4 months-energy restriction-ketogenic intervention arm or a behavioural group intervention and compared with a group of tumor-free normal weight subjects.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Energy restriction-ketogenic intervention (VLCKD)-breast cancer arm (Experimental): Breast cancer patients with obesity will follow an energy-restricted-ketogenic dietary five steps program, which includes lifestyle and behavioral modification support. The first three steps consist of a VLCKD (600 -800 kcal/day), low in carbohydrates (< 50 g daily from vegetables) and lipids (only 10 g of olive oil per day). Throughout these ketogenic phases, supplements of vitamins and minerals supplements, such as K, Na, Mg, Ca, and omega-3 fatty acids will be administered. These three steps will be maintained until the patient lost the target amount of weight, ideally 80%. In steps 4 and 5, the patient started a low-calorie diet (800 -1500 kcal/day) and followed by a maintenance diet that will consist of an eating plan balanced in carbohydrates, protein, and fat (1500 and 2000 kcal/day).
  Interventions: Other: Very low calorie ketogenic diet (VLCKD)
- Group educational intervention program (IGOBE)-breast cancer arm (Experimental): Breast cancer patients with obesity will follow structured program of change of habits that will consist of a balanced hypocaloric diet, following the criteria of both the recommendations from Spanish Society of Study of Obesity (SEEDO) 2007, the American Dietetic Guidelines 2010, the Consensus SEEDO 2012 and the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society Guideline for the Management of Overweight and Obesity in Adults 2014. Coinciding all in pointing out that the hypocaloric diet should represent a deficit of about 500 to 1000 kcal / day with respect to the habitual intake of the patient in question. The intervention group will be included in a structured program of habits change and exercise. In the intensive phase of the intervention patients will assist to 6 additional weekly visits, with 15 patients per group and a duration of 60 minutes each.
  Interventions: Behavioral: Group educational intervention program (IGOBE)
- Energy restriction-ketogenic intervention (VLCKD)-tumor free arm (Experimental): Tumor-free patients with obesity will follow an energy-restricted-ketogenic dietary five steps program, which includes lifestyle and behavioral modification support. The first three steps consist of a VLCKD (600 -800 kcal/day), low in carbohydrates (< 50 g daily from vegetables) and lipids (only 10 g of olive oil per day). Throughout these ketogenic phases, supplements of vitamins and minerals supplements, such as K, Na, Mg, Ca, and omega-3 fatty acids will be administered. These three steps will be maintained until the patient lost the target amount of weight, ideally 80%. In steps 4 and 5, the patient started a low-calorie diet (800 -1500 kcal/day) and followed by a maintenance diet that will consist of an eating plan balanced in carbohydrates, protein, and fat (1500 and 2000 kcal/day).
  Interventions: Other: Very low calorie ketogenic diet (VLCKD)
- Group educational intervention program (IGOBE)-tumor free arm (Experimental): Tumor-free patients with obesity will follow structured program of change of habits that will consist of a balanced hypocaloric diet, following the criteria of both the recommendations from Spanish Society of Study of Obesity (SEEDO) 2007, the American Dietetic Guidelines 2010, the Consensus SEEDO 2012 and the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society Guideline for the Management of Overweight and Obesity in Adults 2014. Coinciding all in pointing out that the hypocaloric diet should represent a deficit of about 500 to 1000 kcal / day with respect to the habitual intake of the patient in question. The intervention group will be included in a structured program of habits change and exercise. In the intensive phase of the intervention patients will assist to 6 additional weekly visits, with 15 patients per group and a duration of 60 minutes each.
  Interventions: Behavioral: Group educational intervention program (IGOBE)
- Non intervention arm-breast cancer arm (No Intervention): This arm will include patients with obesity and normal weight women with breast cancer that will follow the normal clinical practice in their oncological therapy without intervention to lose weight in the group of patients with excess body weight.

INTERVENTIONS:
Other: Very low calorie ketogenic diet (VLCKD) — Weight loss therapies in patients with excess body weight based on a ketogenic diet
  Arms: Energy restriction-ketogenic intervention (VLCKD)-breast cancer arm; Energy restriction-ketogenic intervention (VLCKD)-tumor free arm
Behavioral: Group educational intervention program (IGOBE) — Balanced hypocaloric diet plus structured groupal program of habits change and exercise
  Arms: Group educational intervention program (IGOBE)-breast cancer arm; Group educational intervention program (IGOBE)-tumor free arm

SUMMARY:
Obesity could become the first evitable cause of breast cancer in the near future. Due to the relatively slow rate of development in this field, greater efforts must be applied in this area. The HYPOTHESIS of this work is that "a therapy to lose weight in breast cancer women with obesity during the oncological treatment could contribute to slowing carcinogenesis, and to improve the response to the chemotherapy, survival and prevent future recurrences by erasing deleterious epigenetic marks". A group of breast cancer women with obesity (n=90) will be treated to lose weight during the oncologic treatment with a low calorie-ketogenic diet or a group educational intervention program of healthy lifestyle. The reversibility of the obesity-related breast cancer epigenetic signatures (EPIC array and pyrosequencing) and other molecular features (QRTPCR, ELISA assays) in blood leukocytes and plasma and the progression of disease will be compared with an obesity (n=30) and normalweight (n=30) group under conventional anticancer therapy. A matched-group of tumor-free women (n=60) with obesity will be also treated to lose weight with the same nutritional interventions and compared with tumor-free women with normal weight (n=30) in order to evaluate the potential preventive function of weight loss therapies on cancer-related odds. The outcomes of this project will directly benefit overweight and obese patients from healthcare systems, and also to have an economic value supporting pharmaceutical and food industry companies in the design of innovative treatments, useful biomarkers and preventive tools.

DETAILED DESCRIPTION:
Obesity itself is considered the second leading avoidable cause of cancer, after smoking (Renehan and Soerjomataram, 2016;Islami et al., 2019). The worldwide obesity epidemic has shown no signs of abating, better understanding of the mechanisms underlying obesity-associated cancer is urgently needed with the aim to find new therapeutic targets to counteract the obesity-related cancer in general and breast cancer in particular. The increased morbidity and mortality of obesity-related cancer are mostly attributed to dysfunctional adipose tissue. Therefore, targeting the dysfunction of adipose tissue provides a promising strategy for cancer prevention and therapy.

Breast cancer (BC) is the most common female cancer worldwide and the second common cause of cancer-related death in women. In 2018, around 2 million new cases of BC were diagnosed represented 15% of deaths of the 10 most common cancers (Bray et al., 2018). By 2030 cancer is expected to surpass cardiovascular disease being the prevailing cause of death among all age categories, contributing to a 45% increase in the number of malignancies diagnosis during the next 10 years. This is due to the emergence of the increased prevalence of risk factors, mainly diabesity (diabetes mellitus and obesity) in both developed and developing countries (Christodoulatos et al., 2019).

Risk factors for breast cancer include excess weight and metabolic disorders, which have been linked to a poor prognosis of this disease (Bousquenaud et al., 2018;Kliemann et al., 2019;Le et al., 2019). Thus, the World Cancer Research Fund (WCRF) has concluded that healthy lifestyles may help to prevent up to 70% of cancer cases. These include healthy diet eating, regular physical activity, healthy weight, and avoiding smoking and alcohol drinking (Clinton et al., 2019). Obesity is associated with a greater tumor burden in postmenopausal women diagnosed with breast cancer and with a higher degree of tumor. In addition, obesity and overweight are linked to a worse prognosis and an increase in breast cancer death rate. In fact, recently in a work carried out by our research group (Crujeiras et al., 2012), it was found in a homogeneous population in Spain that the prevalence of obesity among breast cancer patients was significantly higher than the prevalence observed among women of the general Spanish population. This increase in prevalence was especially evident in women with postmenopausal breast cancer (Crujeiras et al., 2012). However, although there is epidemiological evidence of the relationship between obesity and cancer, the molecular mechanisms of this relationship is not well known.

Obesity and cancer mechanisms: Adipose tissue secreted factors, inflammation, oxidative stress, epigenetics.

There are several hypothesis that were proposed to be involved in the relationship between obesity and cancer. Among them, the most of the recent studies are being focused on the effect of the dysfunctional adipose tissue observed in obesity (Cabia et al., 2016). Supporting this hypothesis, a recent work of our research group demonstrated that the obese visceral adipose tissue secretome is able to induce higher proliferation of breast tumor cell lines (Crujeiras et al., 2016).

Moreover, recent studies have shown that tumorigenesis is characterized by important differences in the genetic and epigenetic transformation of the epithelium. This transformation involves, among other processes, modifications in DNA methylation and regulation of intracellular microRNAs (miRNAs) which favor tumor progression and metastasis by silencing tumor suppressor genes. Inflammation seems to play an important role in increasing these epigenetic alterations through the increase in the release of cytokines, reactive oxygen species (ROS) and hypoxia (Murata, 2018).

Alterations in gene expression induced by epigenetic modifications have emerged as an alternative whereby the environment can exert harmful effects on the organism. Thus, there are different factors that have the capacity to activate epigenetic regulation such as dietary factors, physical activity and environmental toxicities. In addition, there is evidence on the association between body weight with differential methylation patterns as well as the effect of increased estrogen levels and inflammation on the epigenetic regulation of genes related to carcinogenesis (Crujeiras et al., 2013).

Therefore, one of the possible mechanisms involved in the association between obesity and breast cancer could be the effect of oxidative stress and inflammation induced by excess adiposity on DNA methylation in breast tissue (Crujeiras et al., 2013;Cabia et al., 2016). In this context, recently, we have described that obesity and menopausal state modulate the methylation pattern of breast tumors (Crujeiras et al., 2017b). These differential profile in methylation was observed in breast tumors and could suggest the existence of a specific molecular subtype of breast cancer induced by excess body weight. Because epigenetic mechanisms are reversible and also the inflammation and oxidative stress induced by the dysfunctional adipose tissue of obesity can be reduced, the outcome of obesity-related breast cancer could be improved by a therapy to lose weight in breast cancer women with obesity.

Weight loss in the treatment of obesity-related cancer The strategies to lose weight were demonstrated to be able to reduce the inflammatory and oxidative stress markers in obese patients. Thus, interventions such as calorie restriction and exercise training, may reduce oxidative stress by increasing antioxidant defences, decreasing fat mass, improving glycaemic control, reducing blood lipids and increasing antioxidant intake from fruits or legumes (Crujeiras et al., 2006;Crujeiras et al., 2007). Hence, calorie restriction alone is able to improve obesity-related oxidative stress by enhancing mitochondrial (Crujeiras et al., 2008a;Crujeiras et al., 2009), and it differentially regulates the expression of oxidative stress and inflammation related genes as well as the gene expression of sirtuins, proteins involved in improving the lifespan (Crujeiras et al., 2008b). Most recently, our group have evidenced that an energy restriction-based weight loss intervention is able to reverse the effects of obesity on the expression of liver tumor-promoting genes in animal models (Izquierdo et al., 2019).

The American Society of Clinical Oncology (ASCO) has highlighted that obesity is one of the most cardinal preventable lifestyle risk factor for cancer mortality (Ligibel et al., 2019). There are clinical and economic benefits associated with identifying individuals who should receive preventative or clinical treatment, and weight loss through lifestyle modification (e.g., proper diet and exercise) may be an effective approach. Due to this, recent years, a number of intervention trial studies for breast cancer survivors aimed at weight loss have been conducted worldwide (Winkels et al., 2017;Ando et al., 2019). There are biologic plausibilities that obesity might be an effect modifier of treatment, but supporting evidence from clinical studies is inconsistent (Renehan et al., 2016). Many trials have evaluated the impact of exercise and weight loss interventions on cardiorespiratory fitness, physical functioning, reductions in fatigue among others, but evidence that demonstrates that lifestyle interventions during active treatment affect cancer outcomes, such as recurrence or mortality or response to treatment is limited (Ligibel et al., 2019).

The current trend for obesity treatment is focused on therapies that induce ketosis such as a very-low calorie ketogenic diet that are able to induce a reduction in fat mass by preserving muscle mass (Moreno et al., 2016;Gomez-Arbelaez et al., 2017) or intermittent fasting (Templeman et al., 2020). Since an oncologic point of view, ketogenic diets (KD) have reported potentially beneficial effects, which were able to prevent malignancies and decrease tumor growth. Some studies have even shown increased patient survival, reduced side effects of cytotoxic treatments and intensified efficacy of cancer therapies (Klement, 2019).

Also, therapies based on a group educational intervention program of healthy lifestyle to lose weight have positive results on reducing fat mass and improving lifestyle habits (Porca et al, Clin Nutr, under review) and currently are among the most promising therapeutic strategies to counteract obesity prevalence.

We propose that the promising weight loss strategies to be evaluated in this study during the active oncologic therapy could be useful to improve the response to oncologic therapy and the prognosis of breast cancer women with obesity by reversing the epigenetic marks of obesity-related breast cancer accompanied by a metabolic state improvement.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Primary, histologically confirmed, incident breast cancer diagnostic

Exclusion Criteria:

* Thyroid disorder,
* Diabetes mellitus,
* Cardiovascular disease,
* cerebrovascular disease
* Obesity induced by other endocrine disorders or drugs,
* Participation in any active weight loss program in the previous 3 months.
* Known or suspected narcotic or alcohol abuse,
* Severe depression or any other psychiatric disease,
* Severe liver failure
* Uncontrolled hypertension,
* Orthostatic hypotension,
* hydroelectrolytic or electrocardiographic alterations
* Prescription of drugs that may alter the lipid or glucose profile.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-10-03 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 4 months
  Changes in body weight induced by the nutritional intervention therapies
Fat mass in kg | 4 months
  Changes in fat mass induced by the nutritional intervention therapies
Fat free mass in kg | 4 months
  Changes in fat free mass induced by the nutritional intervention therapies
Visceral fat mass in kg | 4 months
  Changes in visceral fat mass induced by the nutritional intervention therapies
DNA methylation levels | 4 months
  Changes in the pattern of circulating DNA methylation
Score of quality of life questionnaire | 4 months
  changes in the score of Quality of life associated to the interventions
Score of Sleep Quality questionnaire | 4 months
  Changes in the score of Sleep Quality associated to the interventions
Score of Female Sexual Function Index questionnaire | 4 months
  Changes in the score of Female Sexual Function Index associated to the interventions
Concentration of inflammatory biomarkers | 4 months
  Changes associated to the interventions in plasmatic levels of cytokines quantified using a commercial multiplex enzyme-linked immunosorbent assay (ELISA) kit according to the manufacturer's instructions. The following cytokines were analyzed: April, B cell activator factor (BAFF), cluster of differentiation (CD)163, CD30, Chitanase, glycoprotein (Gp)130, interferon (IFN)-α2, IFN-β, IFN-γ, interleukin (IL)-2, IL-6R, IL-11, IL-12(p40), IL-12(p70), IL-22, IL-26, IL-28A, IL-29, IL-35, matrix metalloproteinase (MMP)1, MMP3, Osteocalcin, Pentraxin-3, tumor necrosis factor receptor (TNF)-R1, TNF-R2, Thymic stromal lymphopoietin (TSLP) and Tweak.
Concentration of Oxidative stress biomarkers | 4 months
  Among the oxidative stress biomarkers, the levels of malondialdehyde (MDA) and total antioxidative power (AOP) and 8-hydroxy-2'-deoxyguanosine (8-OHdG) will be evaluated in serum. MDA and AOP will be quantified using colorimetric assay kits . An enzyme immunoassay kit will be used for the quantification of 8-OHdG in the serum.

SECONDARY OUTCOMES:
Diagnostic of cardiotoxicity | 12 months
  echocardiography, troponin levels, cardiac natriuretic peptides levels
Response to Oncological treatment | 12 months
  Reduction in size of a cancer or not evidence of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ana B Crujeiras, Dr, Principal Investigator — Hospital Clinico Universitario de Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabia B, Andrade S, Carreira MC, Casanueva FF, Crujeiras AB. A role for novel adipose tissue-secreted factors in obesity-related carcinogenesis. Obes Rev. 2016 Apr;17(4):361-76. doi: 10.1111/obr.12377. Epub 2016 Feb 24. PMID 26914773
- [Background] Crujeiras AB, Cabia B, Carreira MC, Amil M, Cueva J, Andrade S, Seoane LM, Pardo M, Sueiro A, Baltar J, Morais T, Monteiro MP, Lopez-Lopez R, Casanueva FF. Secreted factors derived from obese visceral adipose tissue regulate the expression of breast malignant transformation genes. Int J Obes (Lond). 2016 Mar;40(3):514-23. doi: 10.1038/ijo.2015.208. Epub 2015 Oct 26. PMID 26443342
- [Background] Crujeiras AB, Cueva J, Vieito M, Curiel T, Lopez-Lopez R, Pollan M, Casanueva FF. Association of breast cancer and obesity in a homogeneous population from Spain. J Endocrinol Invest. 2012 Jul;35(7):681-5. doi: 10.3275/8370. Epub 2012 Apr 18. PMID 22522745
- [Background] Crujeiras AB, Diaz-Lagares A, Carreira MC, Amil M, Casanueva FF. Oxidative stress associated to dysfunctional adipose tissue: a potential link between obesity, type 2 diabetes mellitus and breast cancer. Free Radic Res. 2013 Apr;47(4):243-56. doi: 10.3109/10715762.2013.772604. Epub 2013 Feb 26. PMID 23409968
- [Background] Crujeiras AB, Diaz-Lagares A, Sandoval J, Milagro FI, Navas-Carretero S, Carreira MC, Gomez A, Hervas D, Monteiro MP, Casanueva FF, Esteller M, Martinez JA. DNA methylation map in circulating leukocytes mirrors subcutaneous adipose tissue methylation pattern: a genome-wide analysis from non-obese and obese patients. Sci Rep. 2017 Feb 17;7:41903. doi: 10.1038/srep41903. PMID 28211912
- [Background] Crujeiras AB, Diaz-Lagares A, Stefansson OA, Macias-Gonzalez M, Sandoval J, Cueva J, Lopez-Lopez R, Moran S, Jonasson JG, Tryggvadottir L, Olafsdottir E, Tinahones FJ, Carreira MC, Casanueva FF, Esteller M. Obesity and menopause modify the epigenomic profile of breast cancer. Endocr Relat Cancer. 2017 Jul;24(7):351-363. doi: 10.1530/ERC-16-0565. Epub 2017 Apr 25. PMID 28442560
- [Background] Gomez-Arbelaez D, Bellido D, Castro AI, Ordonez-Mayan L, Carreira J, Galban C, Martinez-Olmos MA, Crujeiras AB, Sajoux I, Casanueva FF. Body Composition Changes After Very-Low-Calorie Ketogenic Diet in Obesity Evaluated by 3 Standardized Methods. J Clin Endocrinol Metab. 2017 Feb 1;102(2):488-498. doi: 10.1210/jc.2016-2385. PMID 27754807
- [Background] Izquierdo AG, Carreira MC, Amil M, Mosteiro CS, Garcia-Caballero T, Fernandez-Quintela A, Portillo MP, Casanueva FF, Crujeiras AB. An energy restriction-based weight loss intervention is able to reverse the effects of obesity on the expression of liver tumor-promoting genes. FASEB J. 2020 Feb;34(2):2312-2325. doi: 10.1096/fj.201901147RR. Epub 2019 Dec 16. PMID 31908001